CLINICAL TRIAL: NCT01075425
Title: Phase I Study of Belinostat (PXD-101) and Velcade (Bortezomib) in Relapsed or Refractory Acute Leukemia/ Myelodysplastic Syndrome
Brief Title: Belinostat and Bortezomib in Treating Patients With Relapsed or Refractory Acute Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12517; NCI-2010-00127 (Registry Identifier: CTRP); RC2CA148431 (NIH)
Record Dates: First submitted 2010-02-15; First posted 2010-02-25 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Acute Lymphocytic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia
Keywords: leukemia; acute leukemia; chronic myelogenous leukemia; myelodysplastic syndrome; relapsed acute leukemia; refractory acute leukemia; belinostat; bortezomib; Velcade; PXD-101
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — Bortezomib; belinostat; Specimen Handling; Blotting, Western; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive belinostat IV over 30 minutes on days 1-5 and 8-12 and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: belinostat; Other: laboratory biomarker analysis; Genetic: western blotting; Other: pharmacological study; Other: flow cytometry

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: belinostat — Given IV
  Other Names: PXD101
Other: laboratory biomarker analysis — Correlative studies
  Other Names: sample collection
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: flow cytometry — Correlative studies
  Other Names: sample analysis

SUMMARY:
RATIONALE: Belinostat and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving belinostat together with bortezomib may kill more cancer cells. PURPOSE: This phase I trial is studying the side effects and best dose of giving belinostat together with bortezomib in treating patients with relapsed or refractory acute leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the recommended phase II doses for the combination of bortezomib and belinostat in patients with relapsed or refractory acute leukemia (AL), myelodysplasia (MDS), and chronic myelogenous leukemia in blast crisis. SECONDARY OBJECTIVES: I. Determine safety and tolerance and describe the toxicities of the combination. II. To demonstrate adequate methods for the assessment of pharmacodynamic response of leukemia cells from the bone marrow and/or peripheral blood in terms of effects on NF-kB (nuclear RelA by immunofluorescence microscopy), NF-kB dependent proteins XIAP and Bcl-xL, and BIM, and document pharmacodynamic responses observed in the course of this study. III. To document activity of the combination observed in the course of this study. OUTLINE: Patients receive belinostat IV over 30 minutes on days 1-5 and 8-12 and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion

* Relapsed or refractory acute leukemia
* acute myeloid leukemia (AML) other than APL
* acute lymphocytic leukemia (ALL)
* acute leukemia that has evolved from a prior myelodysplastic syndrome - no requirement for prior therapy
* myelodysplastic Syndrome (MDS) - International Prognostic Scoring System (IPSS) intermediate-2 or greater
* chronic myelogenous leukemia with myeloid or lymphoid blast crisis
* WBC =< 50 x 10^9/L; hydroxyurea or leukopheresis may be used prior starting treatment
* Prior allogeneic stem cell transplant is allowed provided that >/= 12 months have elapsed since allogeneic transplant; no graft versus host disease is present; not currently on immunosuppressive therapy
* AST, ALT =< 2.5 x upper limit of normal (ULN)
* Female subject who is post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., oral or injectable hormonal methods; barrier methods such as intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study
* Serum total bilirubin =< 1.5 x upper limit of normal
* Serum potassium >= 3.5 mEq/L and serum magnesium >= 1.7 mEq/dL (electrolytes may be corrected with supplementation)
* ECOG Performance Status (PS) =<2
* Creatinine =< 1.5 x upper limit of normal or calculated or actual creatinine clearance > 45 mL/min

Exclusion

* Willing and medically suitable for remission induction with other agents in anticipation of a potentially curative allogeneic bone marrow transplant
* Known CNS malignant disease
* Prior severe allergic reactions to bortezomib, mannitol, boron, belinostat or compounds of the hydroxamate class or arginine
* Grade 1 with pain or Grade >= 2 peripheral neuropathy or paresthesias within 14 days before enrollment
* History of sustained ventricular tachycardia, ventricular fibrillation, Torsade de Pointes, or resuscitated cardiac arrest

  • History of resuscitated cardiac arrest. Note: persons without pre-existing cardiovascular comorbidities who have experienced resuscitated cardiac arrest in the setting of sepsis ARE eligible provided they have no residual cardiac abnormalities and providing they do not require ongoing medication to manage cardiac issues as an outcome of such an event.
* Conduction abnormality or concomitant treatment with an anti-arrhythmic agent to prevent or control arrhythmia
* Known congenital long QT syndrome
* Clinically significant infection including infection with HIV, or active hepatitis B or C
* Significant cardiovascular disease, hypertrophic cardiomegaly or restrictive cardiomyopathy, myocardial infarction within the past 6 months, unstable angina
* Baseline QTc interval > 450 msec
* Planned or ongoing treatment with any drug that may be risk of causing Torsades de Pointes
* Persistent blood pressure (BP) of >=160/95
* Serious medical or psychiatric illness likely to interfere with patient participation
* Pregnant or nursing
* Diagnosis or treatment for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy
* Planned ongoing treatment with other drugs thought to potentially adversely interact with belinostat
* Strong or moderate CYP3A4 inhibitors
* Patient has received other investigational drugs within 14 days before enrollment
* If steroids for cancer control have been used, patients must be off these agents for >/= 1 week before starting treatment. Exception: maintenance therapy for non-malignant disease with prednisone or steroid equivalent dose < 10 mg/day is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Recommended phase II doses for the combination of bortezomib and belinostat | 2 years

SECONDARY OUTCOMES:
Toxicity | 2 years
Pharmacodynamic response | 2 years
Activity of belinostat and bortezomib | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, Study Chair — Virginia Commonwealth University; Beata Holkova, MD, Principal Investigator — Massey Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/